CLINICAL TRIAL: NCT00189228
Title: Not a Drug Trial. We Are Using Anti-IgE to Examine the Role of Pulmonary Mast Cells in Asthma
Brief Title: Immune Dysfunction in Allergic Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mark Schuyler, Professor of Medicine, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UNMSCOR; R01HL044253 (NIH); NCT00201097 (obsolete NCT alias)
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- xolair (Experimental): This is a single arm, parallel study examining differences of therapeutic outcomes of Xolair. Xolair is being examined as an intervention that might change the outcome of immunization.
  Interventions: Drug: Xolair

INTERVENTIONS:
Drug: Xolair — Patients are administered Xolair

SUMMARY:
We are using anti-IgE to investigate the role of pulmonary mast cells in asthma.

DETAILED DESCRIPTION:
Subjects with mild allergic asthma are examined before, immediately after and 2 months after a course of treatment with anti-IgE. The following are examined: Allergen skin tests, allergen induced asthma, peripheral blood basophils, pulmonary bronchial mucosal mast cells.

ELIGIBILITY:
Inclusion Criteria:

Mild asthma, adults -

Exclusion Criteria:

children. on inhaled or systemic steroids

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schuyler, MD, Study Director — UNM HSC
Locations (1):
- UNM HSC, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from the University community
Pre-assignment Details: No events prior to the study
Groups:
- Xolair: This is not a drug study examining differences of therapeutic outcomes. This is an open label, non randomized single dose level study in which patients will be treated for 85 days with rhuMAB-E25 (Xolair) and followed for a total of 300 days. The dose of Xolair is determined by the patient's total serum IgE and body weight and is administered subcutaneously every 2 or 4 weeks. Outcome is serum anti-KLH antibody (immunoglobulin classes).
Period: Overall Study
Arm/Group | Xolair
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Xolair: This is not a drug study examining differences of therapeutic outcomes. It uses Xolair as an intervention that might change the outcome of immunization.
Arm/Group | Xolair
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Anti-KLH Antibody. This is Measured by ELISA and Expressed as ELISA Units Which Are Derived by Dilution of Serum Samples Until the Result Falls on a Linear Portion of the Response Curve. Final Values Are Derived From ELISA Units and the Serum Dilution
Description: Asthma and control patients are immunized with KLH. Mean levels of anti-KLH antibody as described above. This is measured by ELISA and expressed as ELISA units which are derived by dilution of serum samples until the result falls on a linear portion of the response curve. Final values are derived from ELISA units and the serum dilution
Time Frame: 6 months
Population: Anti-KLH antibody levels of the groups (asthmatics treated with Xolair and placebo) were compared. Both parametric and non parametric statistical techniques were used. There were no differences between the groups.
Measure: Mean (Standard Error); unit: Units of anti-KLH antibody
Arm/Group | Xolair
Number analyzed (Participants) | 18
Units of anti-KLH antibody | 18 (2)
Statistical Analysis 1: Comparison: Xolair; This is not a drug study; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Xolair
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No